CLINICAL TRIAL: NCT05486494
Title: Former Spine Tango Registry Now DWG Registry
Brief Title: Spine Registry University Hospital of Cologne- Department of Orthopedics
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Ayla Yagdiran, Senior Consultant, University of Cologne
Other Study IDs: 09-182
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Outcome, Fatal; Spondylodiscitis; Vertebral Osteomyelitis
Keywords: Quality of Life, Treatment Failure, Relapse, Spondylodiscitis, Vertebral Osteomyelitis
MeSH Terms: conditions — Discitis; Recurrence | interventions — Therapeutics; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment (non- surgical/surgical) — Treatment Outcome based on different aspects

SUMMARY:
Between January 2008 and December 2020 all patients with spine diseases were registered prospectively in the former European Spine Tango registry and later german DWG registry at the department of orthopedics and trauma at the university of cologne.

DETAILED DESCRIPTION:
The following data were prospectively collected after enrollment: age, sex, body mass index (BMI), length of hospital stay, affected spine segment, previous surgical procedures on the spine, conservative or operative treatment including type of surgical treatment and American Society of Anesthesiologists (ASA) Physical Status Classification System.

In addition the following quality of life scores were collected: Oswestry Disability Score (ODI), Core Outcome Measures Index(COMI), Short Form- 36 (SF- 36) and Euroqol- 5D (EQ- 5D).

ELIGIBILITY:
Inclusion Criteria:

* Spine disease

Exclusion Criteria:

* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Within all patients spondylodiscitis/ vertebral osteomyelitis patients were analyzed in detail.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life Data after surgery | 2008- 2020
  Definition of Thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Yagdiran, M.D., Principal Investigator — University of Cologne

IPD SHARING:
Plan to Share IPD: No
none of the data are shared